CLINICAL TRIAL: NCT04779346
Title: Immunity Against Severe Acute Respiratory Syndrome Coronavirus 2 Disease (COVID-19) in the Oncology Outpatient Setting: Prevalence and Serological Immunity in the Oncology Outpatient Clinic of the University Medical Center Hamburg-Eppendorf
Brief Title: Immunity Against Severe Acute Respiratory Syndrome Coronavirus 2 Disease (COVID-19) in the Oncology Outpatient Setting
Acronym: COVIDOUT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-10275-BO-ff
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Cancer; Covid19; Immunity
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatient cancer patients: Cancer patients who are regularly treated in the Oncology Outpatient Clinic of the University Medical Center Hamburg-Eppendorf (UKE)

SUMMARY:
The COVIDOUT study will prospectively investigate the serological immunity of outpatient cancer patients to evaluate the prevalence of previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infections and dependency of serological immunity on systemic (chemo)therapy after COVID19 disease as well as after vaccination.

DETAILED DESCRIPTION:
In this prospective observational study all cancer patients who are regularly treated in the Oncology Outpatient Clinic of the University Medical Center Hamburg-Eppendorf (UKE) will be included in the study upon consent.

Data will be collected as follows:

(i) Serological antibody screening at study inclusion and every 3 months (ia) In case of vaccination monthly screening for 3 months (ii) Routine clinical data: demographic and biometric data, medical history, common laboratory parameters (iii) Patient questionnaire: assessment of past COVID-19 infection, past COVID-19 specific symptoms, social environment, vaccination

Recruitment is limited to a one-year period (December 2020 - December 2021)

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of cancer
* Active disease or (in case of cure) last systemic therapy <12 months
* Signed informed consent

Exclusion Criteria:

* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of cancer patients who are regularly treated in the Oncology Outpatient Clinic of the University Medical Center Hamburg-Eppendorf (UKE)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of SARS-CoV-2 antibody positive patients | 1 year
  Measured in percentage
Rate of SARS-CoV-2 antibody positivity after 3, 6, 9, 12 months in previously SARS-CoV-2 antibody positive patients | Up to 1 year
  Measured in percentage
Rate of SARS-CoV-2 antibody positivity after 3, 6, 9, 12 months in previously SARS-CoV-2 vaccinated patients | Up to 1 year
  Measured in percentage

SECONDARY OUTCOMES:
Rate of unknown prior COVID19 disease in SARS-CoV-2 antibody positive patients | 1 year
  Measured in percentage
Rate of cancer entities in SARS-CoV-2 antibody positive patients | 1 year
  Measured in percentage
Rate of therapy modalities in SARS-CoV-2 antibody positive patients | 1 year
  Measured in percentage
Subgroup analysis of SARS-CoV-2 antibody positivity after 3, 6, 9, 12 months in previously SARS-CoV-2 vaccinated patients | Up to 1 year
  Dependency of rate on cancer entity, therapy modality, age, sex and immune status [Measured in percentage]
Rate of re-infection in SARS-CoV-2 antibody positive patients | 1 year
  Measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Sinn, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data will be shared